CLINICAL TRIAL: NCT00035165
Title: An Open-Label Phase IIa Trial Evaluating the Safety and Efficacy of EPO906 as Therapy in Patients With Advanced Melanoma
Brief Title: EPO906 Therapy in Patients With Advanced Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2206
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Melanoma
Keywords: melanoma; cancer; tumor; tumour; malignant; metastatic; intravenous; epothilone
MeSH Terms: conditions — Melanoma; Neoplasms; Neoplasm Metastasis | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: epothilone b

INTERVENTIONS:
Drug: epothilone b — intravenous 2.5 mg/m2 as a 5 minutes bolus infusion once every week for three weeks followed by one week off
  Other Names: Patupilone, EPO906

SUMMARY:
This study will examine whether the new investigational drug EPO906, given by intravenous infusion (IV directly into the vein), is effective in shrinking tumors and preventing the growth of cells that cause melanoma.

ELIGIBILITY:
Inclusion Criteria

The following patients may be eligible for this study:

* Patients with advanced metastatic melanoma defined as poor prognosis Stage III melanoma and Stage IV disease, which has been histologically or cytologically confirmed with at least one measurable lesion not including bone metastases (if previous radiation treatment, the target lesion must have demonstrated progression since the radiation)
* Patients with poor prognosis Stage III melanoma must have locally advanced unresectable disease that is measurable (repeat histological or cytological confirmation is not necessary at the time of study entry if previous results are available and there is no question in the investigator's opinion as to the diagnosis)
* Must have a life expectancy of greater than three (3) months
* Prior immunotherapy with interferon alpha in the adjuvant setting is permitted, but must have been completed > 4 weeks prior to treatment
* Prior vaccine therapy is permitted, but must have been completed > 4 weeks prior to treatment
* Patient has no major impairment of hematological function (red blood cell transfusions and repeat evaluations for study entry are allowed).

Exclusion Criteria

The following patients are not eligible for this study:

* Patients with choroidal ocular melanoma
* Patients with symptomatic CNS metastases or leptomeningeal involvement
* Patients with renal or hepatic dysfunction
* Patients with any peripheral neuropathy or unresolved diarrhea greater than Grade 1
* Patients with severe cardiac insufficiency
* Patients taking Coumadin or other warfarin-containing agents with the exception of low dose Coumadin (1 mg or less) for the maintenance of in-dwelling lines or ports
* Patients who have received any investigational compound or anti-melanoma vaccine within the past 28 days or those who are planning to receive other investigational drugs while participating in the study
* Patients who had received radiotherapy within the last 4 weeks to a site which will be the reference for disease assessment (however, new or progressive lesions in the previously irradiated fields of these patients may be used for disease assessment and patients must have recovered from the side effects of radiotherapy)
* Patients receiving chemotherapy within the last four weeks
* History of another malignancy within 5 years prior to study entry except curatively treated non-melanoma skin cancer or cervical cancer in situ
* Patients with active or suspected acute or chronic uncontrolled infection including abcesses or fistulae
* HIV+ patients
* Pregnant or lactating females.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-03; Primary Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Tumor response (complete response (CR), partial response (PR), stable disease (SD)) | at screening, at least every eight weeks (one week following the last dose of EPO906 in every even-numbered cycle)
  Objective tumor response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines assessed by radiologic techniques and/or physical examination.

SECONDARY OUTCOMES:
Number and percentage of patients with Adverse events | as necessary
  Safety and tolerabilty of EPO906: Safety assessments consisted of monitoring and recording of all adverse events (AEs) and serious adverse events (SAEs), the regular monitoring of hematology, blood chemistry and urine values, regular measurement of vital signs and the performance status.
Objective response rate (ORR) | at screening, at least every eight weeks (one week following the last dose of EPO906 in every even-numbered cycle)
Time to disease progression (TTP) | at screening, at least every eight weeks (one week following the last dose of EPO906 in every even-numbered cycle)
Overall Survival (OS) | from the date of the first dose of treatment to date of death from any cause, or the last date the patient is known to be alive
Tumor-specific mutations and gene expression changes in tumor cells with blood cells and plasma | prior to the first treatment with EPO906, on the day of any clinically indicated tumor biopsy/resection and on the day of each tumor assessment
  For biomarker development

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - University of Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Comprehensive Cancer Center@ Our Lady if Mercy Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oklahoma Oncology, Inc., Tulsa, Oklahoma
  - UPMC Health Systems, Pittsburgh, Pennsylvania